CLINICAL TRIAL: NCT00640549
Title: Impact of Atorvastatin on the Distribution, Composition, and Metabolism of LDL and HDL Subfractions: A Double-blind Placebo-controlled Phase IV Study With Patients Suffering From Combined Hyperlipidemia and Diabetes. Atorvastatin and LDL Profile in NIDDM (ALPIN Study)
Brief Title: Atorvastatin and LDL Profile in Non-Insulin Dependent Diabetes Mellitus
Acronym: ALPIN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2581040
Record Dates: First submitted 2008-03-14; First posted 2008-03-21 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Hyperlipidemia; Diabetes Mellitus, Type 2; Non-Insulin Dependent Diabetes Mellitus
Keywords: LDL-subfractions, HDL-subfractions, non insulin dependent diabetes mellitus (NIDDM), hyperlipidemia, atorvastatin
MeSH Terms: conditions — Hyperlipidemias; Diabetes Mellitus, Type 2 | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- 1 (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — After a run-in phase of 4 weeks eligible patients were randomized at a ratio of 2 : 1 (atorvastatin : placebo). Patients in the atorvastatin group were treated with atorvastatin 20 mg tablets administered once daily orally for 8 weeks.
  Other Names: Lipitor, Sortis
  Arms: 1
Drug: Placebo — After a run-in phase of 4 weeks eligible patients were randomized at a ratio of 2 : 1 (atorvastatin : placebo). Patients in the placebo group were treated with placebo 20 mg tablets administered once daily orally for 8 weeks.
  Arms: 2

SUMMARY:
The study will investigate the effects of atorvastatin on the concentrations of small, dense LDL and HDL subfractions in patients with diabetes and the underlying mechanisms of these effects.

DETAILED DESCRIPTION:
This study was terminated on October 6, 2004. The study terminated prematurely because of a higher screening failure rate than expected. There were no safety or efficacy reasons involved in the decision to terminate.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with a diagnosis of type 2 diabetes mellitus who either have never had a major adverse cardiac event (MACE) diagnosed before or who had a MACE diagnosed at least 6 months ago, but who, according to the judgement of the treating general practitioner, do not receive any hyperlipidemic therapy. Major adverse cardiac events (MACE) include myocardial infarction, coronary angioplasty, coronary artery bypass graft or other revascularization procedures.

At Screening:

Visit 1 (week -4):

1. Male patients aged >35 and ≤75 years and postmenopausal female patients ≤75 years with a diagnosis of type 2 diabetes mellitus
2. Patients have been euthyroid for at least six months
3. Written informed consent obtained

   At Visit 2 (week 0):
4. LDL cholesterol ≥130 mg/dl (3.3 mmol/l ) and <190 mg/dl (4.9 mmol/l)
5. Triglycerides <150 mg/dl (1.69 mmol/l ) and <600 mg/dl (11.3 mmol/l)
6. Sum of LDL-5 and LDL-6 cholesterol ≥25 mg/dl (0.65 mmol/l)
7. Follicle stimulating Hormone (FSH) >30 U/l in female patients aged <60 years or FSH >20 U/l in female patients aged ≥60 years

Exclusion Criteria:

* HbA1c > 8.0
* Creatine kinase (CK) >5 times the upper limit of normal
* Patients having taken lipid lowering medication within 8 weeks of the screening visit

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2003-03; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Changes in concentration of HDL subfractions 2a and 2b compared with screening (visit 1) | 8 weeks (visit 4)
Changes in concentration of LDL subfractions LDL-5 and LDL-6 compared with screening (visit 1) | 8 weeks (visit 4)

SECONDARY OUTCOMES:
Changes in concentration of apolipoprotein B in VLDL, IDL, LDL-1 through LDL-6 and apolipoprotein A I in HDL subfractions 2a, 2b, and HDL-3 compared with screening (visit 1) | 8 weeks (visit 4)
Changes in Cholesterol ester transfer protein (CETP), lipoprotein and hepatic lipase activity compared with screening (visit 1) | 8 weeks (visit 4)
Changes in concentration of triglycerides, LDL, and HDL compared with screening (visit 1) | 8 weeks (visit 4)
Changes in size of LDL subfractions compared with screening (visit 1) | 8 weeks (visit 4)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Germany (12):
  - Pfizer Investigational Site, BAD Muenster AM Stein
  - Pfizer Investigational Site, Bosenheim
  - Pfizer Investigational Site, Bretten
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Duisburg
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Goch
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Künzing
  - Pfizer Investigational Site, Offenbach
  - Pfizer Investigational Site, Rain
  - Pfizer Investigational Site, Schwabenheim

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581040&StudyName=Atorvastatin%20and%20LDL%20Profile%20in%20Non-Insulin%20Dependent%20Diabetes%20Mellitus%0A